CLINICAL TRIAL: NCT04794101
Title: Phase 3 Follow-up Study of AAV5-hRKp.RPGR for the Treatment of X-linked Retinitis Pigmentosa Associated With Variants in the RPGR Gene
Brief Title: Follow-up Gene Therapy Trial for the Treatment of X-linked Retinitis Pigmentosa Associated With Variants in the RPGR Gene
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MGT-RPGR-022; MGT-RPGR-022 (Other: Janssen Research & Development, LLC); 2020-002255-37 (EudraCT Number); 2024-511411-25-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-12-15; First posted 2021-03-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: X-Linked Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: 97 participants randomized in MGT-RPGR-021. 64 participants randomized to Immediate treatment arm. 33 participants randomized to the deferred arm. These participants will be treated in MGT-RPGR-022. All participants to be followed for 60 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Deferred Treatment From MGT-RPGR-021 of Intermediate Dose (Experimental): Deferred treatment
  Interventions: Biological: Genetic: AAV5-hRKp.RPGR Intermediate Dose
- Already Treated in MGT-RPGR-021 (Experimental): Already treated
  Interventions: Biological: Genetic: AAV5-hRKp.RPGR Intermediate Dose; Biological: Genetic: AAV5-hRKp.RPGR Low Dose
- Deferred Treatment From MGT-RPGR-021 Low Dose (Experimental): Deferred treatment
  Interventions: Biological: Genetic: AAV5-hRKp.RPGR Low Dose

INTERVENTIONS:
Biological: Genetic: AAV5-hRKp.RPGR Intermediate Dose — Bilateral, subretinal administration of AAV5-hRKp.RPGR - deferred treatment group
  Other Names: botaretigene sparoparvovec
  Arms: Already Treated in MGT-RPGR-021; Deferred Treatment From MGT-RPGR-021 of Intermediate Dose
Biological: Genetic: AAV5-hRKp.RPGR Low Dose — Bilateral, subretinal administration of AAV5-hRKp.RPGR - deferred treatment group
  Other Names: botaretigene sparoparvovec
  Arms: Already Treated in MGT-RPGR-021; Deferred Treatment From MGT-RPGR-021 Low Dose

SUMMARY:
A clinical trial of AAV5-hRKp.RPGR vector for participants with X-linked retinitis pigmentosa (XLRP)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 3 years of age or older, has XLRP confirmed by a retinal specialist and has a predicted disease-causing sequence variant in RPGR confirmed by an accredited laboratory.

Exclusion Criteria:

* None

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2029-09-20 (Estimated); Study Completion 2029-12-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Ocular and Non-ocular Adverse Events | Day 1 - Month 60
  Number of participants with ocular and non-ocular adverse events will be assessed.
Number of Participants With Abnormalities in Laboratory Assessments | Day 1 - Month 60
  Number of participants with abnormalities in laboratory assessments will be assessed.
Change From Baseline in Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart Letter Score in Monocular Assessment | From Baseline - Month 60
  Change from baseline in BCVA by ETDRS chart letter score in monocular assessment will be assessed.
Change From Baseline in Low Luminance Visual Acuity by ETDRS Chart Letter Score in Monocular Assessment | From Baseline- Month 60
  Change from baseline in low luminance visual acuity by ETDRS chart letter score in monocular assessment will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (28):
- United States (10):
  - Shiley Eye Institute Jacobs Retina Center, La Jolla, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Stanford Health Care, Palo Alto, California
  - VitreoRetinal Associates, PA, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Univ of Michigan Medical Center, Ann Arbor, Michigan
  - Duke Eye Center, Durham, North Carolina
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Retina Consultants of Houston, Bellaire, Texas
- Ghent University Hospital, Ghent, Belgium
- Hospital For Sick Children, Toronto, Ontario, Canada
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark
- Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris, France
- Hadassah Medical Center, Jerusalem, Israel
- Italy (4):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale San Paolo, Milan
  - Azienda Ospedaliera Univ.- Università Degli studi della Campania - Luigi Vanvitelli, Napoli
  - IRCCS Fondazione G.B. Bietti per lo Studio e la Ricerca in Oftalmologia ONLUS, Rome
- Netherlands (2):
  - VUMC Amsterdam, Amsterdam
  - Radboudumc, Nijmegen
- Hosp Univ Fund Jimenez Diaz, Madrid, Spain
- Switzerland (2):
  - University Hospital Basel, Eye Clinic/Institute of Molecular and Clinical, Basel
  - Universite de Lausanne, Hopital ophtalmique Jules-Gonin, Lausanne
- United Kingdom (4):
  - NHS Lothian, Edinburgh
  - Gartnavel General Hospital, Glasgow
  - St James University Hospital, Leeds
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No